CLINICAL TRIAL: NCT03891511
Title: TMJ Fibrocartilage Detection Using 3D Fat-Suppressed Spoiled Gradient-Echo Magnetic Resonance Imaging
Brief Title: TMJ Fibrocartilage Detection Using MRI
Acronym: WATS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Universidad Mayor (Other); University of Chile (Other)
Responsible Party: Principal Investigator, Gustavo Moncada, Principal investigator, Clinical Professor of Oral Rehabilitation, Universidad de los Andes, Chile
Other Study IDs: UM20-08-2
Record Dates: First submitted 2019-03-19; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: TMJ Disorders; MRI Scans
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human, aged 18-60 years old, female and male, affected with temporo mandibular disorders
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: MRI scann — MRI will be performed in the TMJ of participants affected with TMD
  Other Names: T1 WATS

SUMMARY:
Objective: The aims of this study will be to detect the fibrocartilage layer (FC) of the human temporomandibular joint (TMJ) using 3D SPGR (Spoiled GRASS sequence) (T1 WATS) sequence and to compare these results with those of conventional magnetic resonance imaging (DP, T2 MRI) sequences in patients with temporomandibular disorders (TMD).

DETAILED DESCRIPTION:
This prospective and observational study will focused on analyzing morphological characteristics of the fibrocartilage layer of the TMJ based on the MRI scans of 59 patients. All 118 TMJs of these patients will be suitable for analysis, (range: 18-60 years old), females and males affected by TMD and did not undergo previous TMJ treatment.

ELIGIBILITY:
Inclusion Criteria:

* Internal derangement in theTMJ

Exclusion Criteria:

* Cardiac pacemaker
* Cochlear implant
* Intracranial vascular clips
* Metal particles in the orbit
* Head or face trauma
* Gout
* Generalized osteoarthrosis
* Joint hyperlaxity
* Congenital malformity
* Facial cysts
* Facial tumors
* Previous TMJ surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: participants will be whites, urban, low , medium low and médium socioeconomic level, from Santiago, Chile.
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Presence of the TMJ Fibrocartilage layer | six months
  The fibrocartilage layer will be evaluated dichotomously (absent/present) Patients will be examined using bilateral MRI (Phillips Intera 1,5 T, Sense Flex S Dual Coil) in the sagittal PD-weighted, T2-weighted and T1-weighted WATS, all in the oblique axis of the mandible condyle and with a closed mouth; dynamic gradient-echo at open mouth at 10 mm, 20 mm and 30 mm of the interincisal distance. Additionally, a coronal PD-weighted sequence with the mouth closed will be performed. Of each TMJ will be taken with 8×8 cm FOV and 0.2 cm spacing. All sequences will carried out using the same equipment and on the same day.
Discontinuity of the TMJ FC layer | six months
  The TMJ fibrocartilage layer will be evaluated dichotomously (continuous/discontinuous).
Fibrocartilage Signal Intensity | six month
  Six regions of interest (ROIs) will be measured in the fibrocartilage layer of each TMJ. (anterior 0°, center 45° and posterior 90°), three in the mandibular condyle and three in the temporal fossa. The fibrocartilage signal intensity in each ROI will be expressed as the mean value of intensity units (Osirix).
  All measurements will be made in a simple blinded system by four different observers (ML, MN, CV, GZ) (chi-square test for interobserver agreement: p˂0.05). Measurements will be made separately in the three MRI sequences (length tool, Osirix Imaging software). In all MRI sequences, TMJ will be magnified at a zoom of 3.6. For the T1 WATS sequence, the window width will be set at 90 intensity Units (IU) (all values above +90 Hounsfield Unit (HU) will be white), and the window level was 80 (IU) (all values below +80 HU will be black). All images will be measured and stored in DICOM format., lengt
Thickness of the TMJ fibrocartilage layer | Six months
  The TMJ FC thickness will be measured (curve tool, Osirix) and will expressed in millimeters.
Length of the TMJ fibrocartilage layer | Six moths
  The lenght of the TMJ FC layer will be measured (curve tool, Osirix) and will expressed in millimeters.
Statistical analysis | seven months
  The Shapiro-Wilk test and Levene's test will be performed to assess normality of data distribution and homogeneity of variance of the measurements, respectively.
  To determine the relationship between the presence or absence of fibrocartilage and the different sequences, Fisher's exact test will be used.
  The thickness, length and signal intensity of the fibrocartilage layer will be expressed as a mean value, separated by MRI sequence, and will be analyzed using descriptive statistics.
  SPSS v14.0 for Windows, statistical software will be used to perform data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Moncada, PhD, Principal Investigator — UAndes, Santiago, Chile
Locations (1):
- San Vicente de Paul Centro de Diagnóstico, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No
No IPD included

REFERENCES:
- [Background] Ren YF, Westesson PL, Isberg A. Magnetic resonance imaging of the temporomandibular joint: value of pseudodynamic images. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 Jan;81(1):110-23. doi: 10.1016/s1079-2104(96)80158-2. PMID 8850494
- [Background] Zhang S, Block KT, Frahm J. Magnetic resonance imaging in real time: advances using radial FLASH. J Magn Reson Imaging. 2010 Jan;31(1):101-9. doi: 10.1002/jmri.21987. PMID 19938046
- [Result] Gibbs SJ, Simmons HC 3rd. A protocol for magnetic resonance imaging of the temporomandibular joints. Cranio. 1998 Oct;16(4):236-41. doi: 10.1080/08869634.1998.11746063. PMID 10029751
- [Result] Brady AP, McDevitt L, Stack JP, Downey D. A technique for magnetic resonance imaging of the temporomandibular joint. Clin Radiol. 1993 Feb;47(2):127-33. doi: 10.1016/s0009-9260(05)81189-4. PMID 8435960
- [Result] Eberhard D, Bantleon HP, Steger W. Functional magnetic resonance imaging of temporomandibular joint disorders. Eur J Orthod. 2000 Oct;22(5):489-97. doi: 10.1093/ejo/22.5.489. PMID 11105405
- [Result] Disler DG, McCauley TR, Wirth CR, Fuchs MD. Detection of knee hyaline cartilage defects using fat-suppressed three-dimensional spoiled gradient-echo MR imaging: comparison with standard MR imaging and correlation with arthroscopy. AJR Am J Roentgenol. 1995 Aug;165(2):377-82. doi: 10.2214/ajr.165.2.7618561.
- [Result] Disler DG, McCauley TR, Kelman CG, Fuchs MD, Ratner LM, Wirth CR, Hospodar PP. Fat-suppressed three-dimensional spoiled gradient-echo MR imaging of hyaline cartilage defects in the knee: comparison with standard MR imaging and arthroscopy. AJR Am J Roentgenol. 1996 Jul;167(1):127-32. doi: 10.2214/ajr.167.1.8659356.
- [Result] Recht MP, Kramer J, Marcelis S, Pathria MN, Trudell D, Haghighi P, Sartoris DJ, Resnick D. Abnormalities of articular cartilage in the knee: analysis of available MR techniques. Radiology. 1993 May;187(2):473-8. doi: 10.1148/radiology.187.2.8475293.
- [Result] Moncada G, Cortes D, Millas R, Marholz C. Relationship between disk position and degenerative bone changes in temporomandibular joints of young subjects with TMD. An MRI study. J Clin Pediatr Dent. 2014 Spring;38(3):269-76. doi: 10.17796/jcpd.38.3.w43m8474433n7ur2. PMID 25095324
- [Result] Dias IM, Coelho PR, Picorelli Assis NM, Pereira Leite FP, Devito KL. Evaluation of the correlation between disc displacements and degenerative bone changes of the temporomandibular joint by means of magnetic resonance images. Int J Oral Maxillofac Surg. 2012 Sep;41(9):1051-7. doi: 10.1016/j.ijom.2012.03.005. Epub 2012 Mar 31. PMID 22464851
- [Result] Larheim TA. Role of magnetic resonance imaging in the clinical diagnosis of the temporomandibular joint. Cells Tissues Organs. 2005;180(1):6-21. doi: 10.1159/000086194. PMID 16088129
- [Result] Tanaka E, Detamore MS, Mercuri LG. Degenerative disorders of the temporomandibular joint: etiology, diagnosis, and treatment. J Dent Res. 2008 Apr;87(4):296-307. doi: 10.1177/154405910808700406. PMID 18362309
- [Result] Stegenga B. Osteoarthritis of the temporomandibular joint organ and its relationship to disc displacement. J Orofac Pain. 2001 Summer;15(3):193-205. PMID 11575190
- [Result] Campos MI, Campos PS, Cangussu MC, Guimaraes RC, Line SR. Analysis of magnetic resonance imaging characteristics and pain in temporomandibular joints with and without degenerative changes of the condyle. Int J Oral Maxillofac Surg. 2008 Jun;37(6):529-34. doi: 10.1016/j.ijom.2008.02.011. Epub 2008 Apr 28. PMID 18440778
- [Result] Kurita H, Kojima Y, Nakatsuka A, Koike T, Kobayashi H, Kurashina K. Relationship between temporomandibular joint (TMJ)-related pain and morphological changes of the TMJ condyle in patients with temporomandibular disorders. Dentomaxillofac Radiol. 2004 Sep;33(5):329-33. doi: 10.1259/dmfr/13269559. PMID 15585811
- [Result] Hauger O, Dumont E, Chateil JF, Moinard M, Diard F. Water excitation as an alternative to fat saturation in MR imaging: preliminary results in musculoskeletal imaging. Radiology. 2002 Sep;224(3):657-63. doi: 10.1148/radiol.2243011227. PMID 12202695
- [Result] Zhang S, Uecker M, Voit D, Merboldt KD, Frahm J. Real-time cardiovascular magnetic resonance at high temporal resolution: radial FLASH with nonlinear inverse reconstruction. J Cardiovasc Magn Reson. 2010 Jul 8;12(1):39. doi: 10.1186/1532-429X-12-39. PMID 20615228
- [Result] Li X, Ma BC, Bolbos RI, Stahl R, Lozano J, Zuo J, Lin K, Link TM, Safran M, Majumdar S. Quantitative assessment of bone marrow edema-like lesion and overlying cartilage in knees with osteoarthritis and anterior cruciate ligament tear using MR imaging and spectroscopic imaging at 3 Tesla. J Magn Reson Imaging. 2008 Aug;28(2):453-61. doi: 10.1002/jmri.21437. PMID 18666183
- [Result] Duc SR, Pfirrmann CW, Schmid MR, Zanetti M, Koch PP, Kalberer F, Hodler J. Articular cartilage defects detected with 3D water-excitation true FISP: prospective comparison with sequences commonly used for knee imaging. Radiology. 2007 Oct;245(1):216-23. doi: 10.1148/radiol.2451060990. Epub 2007 Aug 23. PMID 17717327
- [Result] Dunn TC, Lu Y, Jin H, Ries MD, Majumdar S. T2 relaxation time of cartilage at MR imaging: comparison with severity of knee osteoarthritis. Radiology. 2004 Aug;232(2):592-8. doi: 10.1148/radiol.2322030976. Epub 2004 Jun 23. PMID 15215540
- [Result] Guler N, Yatmaz PI, Ataoglu H, Emlik D, Uckan S. Temporomandibular internal derangement: correlation of MRI findings with clinical symptoms of pain and joint sounds in patients with bruxing behaviour. Dentomaxillofac Radiol. 2003 Sep;32(5):304-10. doi: 10.1259/dmfr/24534480. PMID 14709605
- [Result] Khan HA, Ahad H, Sharma P, Bajaj P, Hassan N, Kamal Y. Correlation between magnetic resonance imaging and arthroscopic findings in the knee joint. Trauma Mon. 2015 Feb;20(1):e18635. doi: 10.5812/traumamon.18635. Epub 2015 Jan 7. PMID 25825695
- [Result] Recht MP, Piraino DW, Paletta GA, Schils JP, Belhobek GH. Accuracy of fat-suppressed three-dimensional spoiled gradient-echo FLASH MR imaging in the detection of patellofemoral articular cartilage abnormalities. Radiology. 1996 Jan;198(1):209-12. doi: 10.1148/radiology.198.1.8539380.
- [Result] Wang Y, Wluka AE, Jones G, Ding C, Cicuttini FM. Use magnetic resonance imaging to assess articular cartilage. Ther Adv Musculoskelet Dis. 2012 Apr;4(2):77-97. doi: 10.1177/1759720X11431005. PMID 22870497
- [Result] Welsch GH, Mamisch TC, Weber M, Horger W, Bohndorf K, Trattnig S. High-resolution morphological and biochemical imaging of articular cartilage of the ankle joint at 3.0 T using a new dedicated phased array coil: in vivo reproducibility study. Skeletal Radiol. 2008 Jun;37(6):519-26. doi: 10.1007/s00256-008-0474-z. PMID 18408924
- [Result] Trattnig S, Breitenseher MJ, Huber M, Zettl R, Rottmann B, Haller J, Imhof H. [Determination of cartilage thickness in the ankle joint. an MRT (1.5)-anatomical comparative study]. Rofo. 1997 Apr;166(4):303-6. doi: 10.1055/s-2007-1015429. German. PMID 9198493
- [Result] Siepmann DB, McGovern J, Brittain JH, Reeder SB. High-resolution 3D cartilage imaging with IDEAL SPGR at 3 T. AJR Am J Roentgenol. 2007 Dec;189(6):1510-5. doi: 10.2214/AJR.07.2661. PMID 18029893
- [Result] Hoemann CD, Lafantaisie-Favreau CH, Lascau-Coman V, Chen G, Guzman-Morales J. The cartilage-bone interface. J Knee Surg. 2012 May;25(2):85-97. doi: 10.1055/s-0032-1319782. PMID 22928426
- [Result] Kuroda S, Tanimoto K, Izawa T, Fujihara S, Koolstra JH, Tanaka E. Biomechanical and biochemical characteristics of the mandibular condylar cartilage. Osteoarthritis Cartilage. 2009 Nov;17(11):1408-15. doi: 10.1016/j.joca.2009.04.025. Epub 2009 May 18. PMID 19477310
- [Result] Brem MH, Pauser J, Yoshioka H, Brenning A, Stratmann J, Hennig FF, Kikinis R, Duryea J, Winalski CS, Lang P. Longitudinal in vivo reproducibility of cartilage volume and surface in osteoarthritis of the knee. Skeletal Radiol. 2007 Apr;36(4):315-20. doi: 10.1007/s00256-006-0208-z. Epub 2007 Jan 12. PMID 17219231
- [Result] Mosher TJ, Smith HE, Collins C, Liu Y, Hancy J, Dardzinski BJ, Smith MB. Change in knee cartilage T2 at MR imaging after running: a feasibility study. Radiology. 2005 Jan;234(1):245-9. doi: 10.1148/radiol.2341040041. Epub 2004 Nov 18. PMID 15550376
- [Result] Suenaga S, Ogura T, Matsuda T, Noikura T. Severity of synovium and bone marrow abnormalities of the temporomandibular joint in early rheumatoid arthritis: role of gadolinium-enhanced fat-suppressed T1-weighted spin echo MRI. J Comput Assist Tomogr. 2000 May-Jun;24(3):461-5. doi: 10.1097/00004728-200005000-00020. PMID 10864087